CLINICAL TRIAL: NCT03599544
Title: A Paradigm Sift: Rehabilitation Robotics, Cognitive Skills Training and Function
Brief Title: Rehabilitation Robotics, Cognitive Skills Training and Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was halted prematurely and will not resume due to loss of funding and access to rehabilitation exoskeleton robot (ArmeoSpring), prohibiting completion of project as planned.
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Principal Investigator, Susan Fasoli, ScD OTR/L, Associate Professor, MGH Institute of Health Professions, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P001182; AOTFIRG18FASOLI (Other Grant/Funding Number: American Occupational Therapy Foundation)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: Upper limb function; Arm and hand weakness
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator(s) will be blinded to assigned study group and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robot-Assisted Therapy (RT) (Active Comparator): Armeo & Amadeo robot-assisted intensive upper limb therapy 1 hour sessions 3x week for 6 weeks.
  Interventions: Behavioral: Robot-Assisted Therapy (RT)
- Robot + Active Learning Program(RT-ALPS) (Experimental): Armeo & Amadeo robot-assisted intensive upper limb therapy 1 hour sessions 3x week for 6 weeks plus training in active problem solving, analysis of performance, and goal-setting focused on the transfer of acquired motor skills to daily activities in the home and community.
  Interventions: Behavioral: Robot + Active Learning Program(RT-ALPS)

INTERVENTIONS:
Behavioral: Robot-Assisted Therapy (RT) — Highly intensive robot-assisted therapy for the paretic arm with the Armeo exoskeleton (1 hour sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo robot (3x week for 3 weeks).
  Arms: Robot-Assisted Therapy (RT)
Behavioral: Robot + Active Learning Program(RT-ALPS) — Highly intensive robot-assisted therapy for the paretic arm with the Armeo exoskeleton (1 hour sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo robot (3x week for 3 weeks). In addition, participants will receive training in active problem solving, analysis of performance and goal setting focused on home action plan activities to assist with carry-over and generalization to every day activities.
  Arms: Robot + Active Learning Program(RT-ALPS)

SUMMARY:
This study evaluates the effects of robot-assisted therapy for adults more than 6 months after stroke on upper limb functioning. Half of the participants will receive robot-assisted therapy for the arm affected by stroke, and the other half will receive robot-assisted therapy plus training in how to use the weaker arm during every day activities.

DETAILED DESCRIPTION:
Research has shown that robot-assisted therapy can help people regain control of simple reaching or grasping movements, but these improvements don't generalize well to use of the weaker limb during everyday tasks.

This study aims to refine and test a protocol named the Active Learning Program for Stroke (ALPS), which teaches people to use active problem solving strategies and a home program to improve function. Therapist-delivered ALPS instruction may incorporate use of strategies (e.g. STOP, THINK, DO, CHECK) modeled after the Cognitive Orientation for daily Occupational Performance (CO-OP) approach to improve real-world use of the paretic upper limb. We will evaluate whether the combination of robot-assisted therapy and ALPS training leads to better satisfaction and functional use of the weaker arm in persons with motor impairments more than 6 months after stroke, as compared to robot-assisted therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unilateral stroke more than 6 months prior to study enrollment.
* Stroke type will include both ischemic and hemorrhagic stroke.
* Moderate UE hemiparesis (characterized by initial scores on upper limb subtest of the Fugl-Meyer Assessment (FMA) between 19-47/60)
* Intact cognitive function to understand and actively engage in the ALPS robotic therapy procedures (Montreal Cognitive Assessment Score >/=26/30)during the initial evaluation visit

Exclusion Criteria:

* No more than moderate impairments in paretic UE sensation, passive range of motion, and pain that would limit ability to engage in therapy, as indicated by subtests of the Fugl-Meyer Assessment (FMA) [13]
* Increased muscle tone as indicated by score of >/= 3 on the Modified Ashworth Scale [15];
* Hemispatial neglect or visual field loss measured by the symbol cancellation subtest on the Cognitive Linguistic Quick Test [16]
* Aphasia sufficient to limit comprehension and completion of the treatment protocol
* Currently enrolled or has plans to enroll in other upper limb therapy/research during the study period
* Treatment with Botox injections for the affected arm within the previous 4 months or planned Botox injections before the end of the study
* Contraindications for robot-assisted therapy including recent fracture or skin lesion of paretic UE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Fugl-Meyer Assessment (FMA) at 6 weeks | Baseline and 6 weeks
  The Fugl-Meyer Assessment (FMA) will examine changes in motor function in the paretic upper extremity (UE) during basic reaching and grasping motions. All items are rated by a 3-point ordinal scale (0=cannot perform; 2=performs fully) with a total possible score of 60 points (reflex items will not be administered). Higher scores indicate better performance.
Change from Baseline Motor Activity Log (MAL) Amount of Use (AOU) at 6 weeks | Baseline and 6 weeks
  The Motor Activity Log (MAL) is a self-report measure in which the person is asked to rate their use of the paretic arm and hand during 28 daily activities. Two scales are used for scoring: Amount of Use (AOU) and Quality of Movement (QOM). Scores range from 0 to 5 (0=not used at all, 5=as well as before stroke) and the average score for each scale is used to assess upper limb function. Higher scores indicate better performance.
Change from Baseline Motor Activity Log (MAL) Quality of Movement (QOM) at 6 weeks | Baseline and 6 weeks
  The Motor Activity Log (MAL) is a self-report measure in which the person is asked to rate their use of the paretic arm and hand during 28 daily activities. Two scales are used for scoring: Amount of Use (AOU) and Quality of Movement (QOM). Scores range from 0 to 5 (0=not used at all, 5=as well as before stroke) and the average score for each scale is used to assess upper limb function. Higher scores indicate better performance.
Change from Baseline Fugl-Meyer Assessment (FMA) at 10 weeks | Baseline and 10 weeks
  The Fugl-Meyer Assessment (FMA) will examine changes in motor function in the paretic upper extremity (UE) during basic reaching and grasping motions. All items are rated by a 3-point ordinal scale (0=cannot perform; 2=performs fully) with a total possible score of 60 points (reflex items will not be administered). Higher scores indicate better performance.
Change from Baseline Motor Activity Log (MAL) Amount of Use (AOU) at 10 weeks | Baseline and 10 weeks
  The Motor Activity Log (MAL) is a self-report measure in which the person is asked to rate their use of the paretic arm and hand during 28 daily activities. Two scales are used for scoring: Amount of Use (AOU) and Quality of Movement (QOM). Scores range from 0 to 5 (0=not used at all, 5=as well as before stroke) and the average score for each scale is used to assess upper limb function. Higher scores indicate better performance.
Change from Baseline Motor Activity Log (MAL) Quality of Movement (QOM) at 10 weeks | Baseline and 10 weeks
  The Motor Activity Log (MAL) is a self-report measure in which the person is asked to rate their use of the paretic arm and hand during 28 daily activities. Two scales are used for scoring: Amount of Use (AOU) and Quality of Movement (QOM). Scores range from 0 to 5 (0=not used at all, 5=as well as before stroke) and the average score for each scale is used to assess upper limb function. Higher scores indicate better performance.

SECONDARY OUTCOMES:
Change from Baseline Modified Ashworth Scale (MAS) at 6 weeks | Baseline and 6 weeks
  The Modified Ashworth Scale (MAS) measures velocity-dependent resistance or spasticity during passive range of motion of nine upper limb movements of the weaker arm, using an ordinal scale that ranges from 0 to 4 (0=no increase in muscle tone, 4=affected part rigid in flexion or extension). Lower scores indicate better performance.
Change from Baseline Wolf Motor Function Test (WMFT) Time at 6 weeks | Baseline and 6 weeks
  The Wolf Motor Function Test (WMFT) quantifies motor ability in the paretic arm and hand during functionally based upper limb tasks. It consists of 3 parts that are scored separately: timed performance, strength, and an ordinal Functional Ability Scale (FAS). The FAS is scored by the evaluator post testing on a 6-point ordinal scale from 0 (does not attempt with the involved arm) to 5 (arm does participate; movement appears normal) and timed tasks have a maximum allotted time of 120 seconds. Higher FAS scores, greater grip strength (measured in kg) and faster time to accomplish tasks indicate better performance.
Change from Baseline Wolf Motor Function Test (WMFT) Strength (kg) at 6 weeks | Baseline and 6 weeks
  The Wolf Motor Function Test (WMFT) quantifies motor ability in the paretic arm and hand during functionally based upper limb tasks. It consists of 3 parts that are scored separately: timed performance, strength, and an ordinal Functional Ability Scale (FAS). The FAS is scored by the evaluator post testing on a 6-point ordinal scale from 0 (does not attempt with the involved arm) to 5 (arm does participate; movement appears normal) and timed tasks have a maximum allotted time of 120 seconds. Higher FAS scores, greater grip strength (measured in kg) and faster time to accomplish tasks indicate better performance.
Change from Baseline Wolf Motor Function Test (WMFT) Functional Ability Score (FAS) at 6 weeks | Baseline and 6 weeks
  The Wolf Motor Function Test (WMFT) quantifies motor ability in the paretic arm and hand during functionally based upper limb tasks. It consists of 3 parts that are scored separately: timed performance, strength, and an ordinal Functional Ability Scale (FAS). The FAS is scored by the evaluator post testing on a 6-point ordinal scale from 0 (does not attempt with the involved arm) to 5 (arm does participate; movement appears normal) and timed tasks have a maximum allotted time of 120 seconds. Higher FAS scores, greater grip strength (measured in kg) and faster time to accomplish tasks indicate better performance.
Change from Baseline Canadian Occupational Performance Measure (COPM) at 6 weeks | Baseline and 6 weeks
  The Canadian Occupational Performance Measure (COPM) is a self-report measure to assess upper limb performance during valued daily activities. A Likert scale (Scored from low [1] to high [10]) is used to rate participant performance of selected functional activities. Higher scores indicate better performance.
Change from Baseline Stroke Impact Scale (SIS) at 6 weeks | Baseline and 6 weeks
  The Stroke Impact Scale (SIS) is a disease specific 59-item measure divided into 8 domains: strength, hand function, activities of daily living (ADL)/instrumental activities of daily living (IADL), mobility, communication, emotion, memory and thinking, and participation/role function. Each item is scored on a 5-point Likert-scale from 1 (unable, extremely difficult) to 5 (not difficult at all). Higher scores for each domain indicate better performance.
Change from Baseline Confidence in Arm and Hand Movement (CAHM) Scale at 6 weeks | Baseline and 6 weeks
  The Confidence in Arm and Hand Movement (CAHM) Scale is a self-report measure of upper limb functional use during a variety of functional tasks (e.g. cutting food with knife and fork at restaurant, using potholders to remove a hot casserole from the oven). Participants rate how confident/certain they are that they can successfully complete each task (n=20) on a scale from 0 (very uncertain) to 100 (very certain). Item scores are averaged to provide a total confidence score (Max score = 100 points).
Change from Baseline Home-based Accelerometry: Wearable Sensors at 6 weeks | Baseline and 6 weeks
  The GENEActiv (http://geneactiv.org) wearable sensor is a multi-directional, waterproof sensor used to quantitatively measure upper limb activity during every day living situations. Sensors will be worn on both wrists for 72 hour periods at each assessment point to compare movements of the paretic and intact upper limb during daily activities. A variety of measures (e.g. amount of arm use, ratio of use between both arms) will be derived from the raw data collected from the sensors.
Change from Baseline Modified Ashworth Scale (MAS) at 10 weeks | Baseline and 10 weeks
  The Modified Ashworth Scale (MAS) measures velocity-dependent resistance or spasticity during passive range of motion of nine upper limb movements of the weaker arm, using an ordinal scale that ranges from 0 to 4 (0=no increase in muscle tone, 4=affected part rigid in flexion or extension). Lower scores indicate better performance.
Change from Baseline Wolf Motor Function Test (WMFT) Time at 10 weeks | Baseline and 10 weeks
  The Wolf Motor Function Test (WMFT) quantifies motor ability in the paretic arm and hand during functionally based upper limb tasks. It consists of 3 parts that are scored separately: timed performance, strength, and an ordinal Functional Ability Scale (FAS). The FAS is scored by the evaluator post testing on a 6-point ordinal scale from 0 (does not attempt with the involved arm) to 5 (arm does participate; movement appears normal) and timed tasks have a maximum allotted time of 120 seconds. Higher FAS scores, greater grip strength (measured in kg) and faster time to accomplish tasks indicate better performance.
Change from Baseline Wolf Motor Function Test (WMFT) Strength (kg) at 10 weeks | Baseline and 10 weeks
  The Wolf Motor Function Test (WMFT) quantifies motor ability in the paretic arm and hand during functionally based upper limb tasks. It consists of 3 parts that are scored separately: timed performance, strength, and an ordinal Functional Ability Scale (FAS). The FAS is scored by the evaluator post testing on a 6-point ordinal scale from 0 (does not attempt with the involved arm) to 5 (arm does participate; movement appears normal) and timed tasks have a maximum allotted time of 120 seconds. Higher FAS scores, greater grip strength (measured in kg) and faster time to accomplish tasks indicate better performance.
Change from Baseline Wolf Motor Function Test (WMFT) Functional Ability Score (FAS) at 10 weeks | Baseline and 10 weeks
  The Wolf Motor Function Test (WMFT) quantifies motor ability in the paretic arm and hand during functionally based upper limb tasks. It consists of 3 parts that are scored separately: timed performance, strength, and an ordinal Functional Ability Scale (FAS). The FAS is scored by the evaluator post testing on a 6-point ordinal scale from 0 (does not attempt with the involved arm) to 5 (arm does participate; movement appears normal) and timed tasks have a maximum allotted time of 120 seconds. Higher FAS scores, greater grip strength (measured in kg) and faster time to accomplish tasks indicate better performance.
Change from Baseline Canadian Occupational Performance Measure (COPM) at 10 weeks | Baseline and 10 weeks
  The Canadian Occupational Performance Measure (COPM) is a self-report measure to assess upper limb performance during valued daily activities. A Likert scale (Scored from low [1] to high [10]) is used to rate participant performance of selected functional activities. Higher scores indicate better performance.
Change from Baseline Stroke Impact Scale (SIS) at 10 weeks | Baseline and 10 weeks
  The Stroke Impact Scale (SIS) is a disease specific 59-item measure divided into 8 domains: strength, hand function, activities of daily living (ADL)/instrumental activities of daily living (IADL), mobility, communication, emotion, memory and thinking, and participation/role function. Each item is scored on a 5-point Likert-scale from 1 (unable, extremely difficult) to 5 (not difficult at all). Higher scores for each domain indicate better performance.
Change from Baseline Confidence in Arm and Hand Movement (CAHM) Scale at 10 weeks | Baseline and 10 weeks
  The Confidence in Arm and Hand Movement (CAHM) Scale is a self-report measure of upper limb functional use during a variety of functional tasks (e.g. cutting food with knife and fork at restaurant, using potholders to remove a hot casserole from the oven). Participants rate how confident/certain they are that they can successfully complete each task (n=20) on a scale from 0 (very uncertain) to 100 (very certain). Item scores are averaged to provide a total confidence score (Max score = 100 points).
Change from Baseline Home-based Accelerometry: Wearable Sensors at 10 weeks | Baseline and 10 weeks
  The GENEActiv (http://geneactiv.org) wearable sensor is a multi-directional, waterproof sensor used to quantitatively measure upper limb activity during every day living situations. Sensors will be worn on both wrists for 72 hour periods at each assessment point to compare movements of the paretic and intact upper limb during daily activities. A variety of measures (e.g. amount of arm use, ratio of use between both arms) will be derived from the raw data collected from the sensors.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Study Chair — Spaulding Rehabilitation Hospital
Locations (2):
- United States (2):
  - MGH Institute of Health Professions, Boston, Massachusetts
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No